CLINICAL TRIAL: NCT02476968
Title: An Open Label, Single Arm, Multicentre Study to Assess the Clinical Effectiveness and Safety of Lynparza (Olaparib) Capsules Maintenance Monotherapy in Platinum Sensitive Relapsed Somatic or Germline BRCA Mutated Ovarian Cancer Patients Who Are in Complete or Partial Response Following Platinum Based Chemotherapy (ORZORA).
Brief Title: To Assess the Efficacy and Safety of Olaparib Maintenance Monotherapy in the Treatment of Ovarian Cancer
Acronym: ORZORA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D0816C00012
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: BRCA or HRR+ Mutated Ovarian Cancer Patients
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaparib (Other): Open Label Drug
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib Capsule - 50 mg. Olaparib capsules will be packed in high-density polyethylene (HDPE) bottles with child-resistant closures. Each bottle will contain 120 capsules and 4 bottles will be dispensed for a 4 weekly visit, with a 2 day overage.
  Patients will be administered olaparib capsules orally at a dose of 400 mg twice daily.
  Eight 50 mg olaparib capsules should be taken at the same time each day approximately 12 hours apart with approximately 240 mL of water.
  Other Names: Lynparza

SUMMARY:
This is a prospective, open-label, single arm, multi-center study to assess the real world clinical effectiveness and safety of olaparib maintenance monotherapy as the capsule formulation (in line with the EU approved prescribing information) and will be conducted in platinum-sensitive relapsed high grade epithelial ovarian cancer patients (including patients with primary peritoneal and / or fallopian tube cancer) who carry germline or somatic BRCA mutations (documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious [known or predicted to be detrimental/lead to loss of function]).

DETAILED DESCRIPTION:
The study will recruit approximately 250 patients with sBRCAm disease or gBRCAm disease, with the aim to accrue a minimum of 50 patients with sBRCAm disease.

Patients with an unknown germline BRCA mutated status or gBRCAwt disease or previously identified as having a BRCAm disease by a tumour test will be considered for screening and will undergo, upon informed consent signature, central tumor and blood testing to determine their BRCA mutation status. In addition to central BRCA testing, patients screened for the study with unknown BRCA status or with known gBRCAwt status, for whom an adequate archival tumour tissue sample is available, will be tested for qualifying HRR gene alterations. Patients confirmed to carry a deleterious or suspected deleterious BRCA-independent genetic alteration in any of 13 genes involved in the Homologous Recombination Repair (HRR) pathway (HRRm cohort) will be allowed into an additional exploratory cohort (HRRm cohort). It is expected that approximately 25 patients will be included in the HRRm cohort before the target number of 250 patients with BRCAm disease is reached.

Patients will be assigned olaparib capsules orally 400 mg twice daily. They should initiate olaparib treatment within 8 weeks after their last dose of platinum-containing chemotherapy (last dose is the day of the last infusion) and will be assessed every 4 weeks whilst on treatment.

All patients will have clinical and objective radiological tumour assessments according to modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines at baseline and every 12 weeks relative to date of enrolment, until objective radiological disease progression as determined by the investigator. Patients could continue to receive olaparib for as long as determined by the investigator, until objective radiological disease progression or as long as in the investigator's opinion they are benefiting from treatment in relation to other clinical assessments and they do not meet any other discontinuation criteria. Once a patient has discontinued olaparib she will be managed as per local clinical practice but will remain in the study and data will be collected on subsequent treatments, progression, overall survival and safety.

For exploratory analysis purposes, patients will be asked to provide consent to:

1. Optional tumour samples at baseline and at disease progression
2. An optional blood sample only for patients with a confirmed sBRCAm or HRRm disease

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Age 18 years or over
3. Documented germline or somatic mutation in BRCA1 or BRCA2 genes that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function) [Genetic counselling for patients with germline BRCA mutations should be performed according to local regulations] Or Tumour BRCAwt status and documented qualifying mutation in any of 13 genes involved in the HRR pathway, excluding BRCA1 and BRCA2 (ATM, BARD1, BRIP1,CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D,and RAD54L), identified by the Lynparza HRR Assay in archival tumour tissue (i.e.,BRCA-independent HRRm)
4. Patients with platinum sensitive relapsed high grade epithelial ovarian cancers (including primary peritoneal and/or fallopian tube cancer):

   - Platinum sensitive disease is defined as disease progression ≥6 months after completion of their last dose of platinum based chemotherapy
5. Patients should have received at least 2 previous lines of platinum containing therapy prior to enrolment:

   - For the last chemotherapy course immediately prior to enrolment on the study, patients must be, in the opinion of the investigator, in response (partial or complete radiological response) and no evidence of a rising CA-125, following completion of this chemotherapy course.
6. Patients must have normal organ and bone marrow function measured within 28 days of enrolment, as defined below:

   * Haemoglobin ≥ 10.0 g/dL with no blood transfusions in the past 28 days
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
7. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase [SGOT]) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase [SGPT]) ≤ 2.5 x institutional ULN unless liver metastases are present in which case they must be ≤ 5x ULN
8. Creatinine clearance > 50 ml/min (calculated)
9. Patients must be postmenopausal or have evidence of non-childbearing status for women of childbearing potential.

Postmenopausal is defined as any of the following:

* Amenorrhoea for 1 year or more following cessation of exogenous hormonal treatments
* For women under 50 years old, luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range
* Radiation-induced oophorectomy, with interval of 1 year or more since last menses
* Chemotherapy-induced menopause, with interval of 1 year or more since last menses
* Surgical sterilisation (bilateral oophorectomy or hysterectomy).

Exclusion Criteria:

1. Patients previously diagnosed with gBRCAm disease
2. Participation in another clinical study with an investigational product during the most recent chemotherapy course
3. Patients with a known hypersensitivity to olaparib or any of the excipients of the product
4. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) or major surgery within 3 weeks prior to olaparib treatment. Major surgery within 3 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
5. Persistent toxicities Common Terminology Criteria for Adverse Event (CTCAE) grade 2 caused by previous cancer therapy, excluding alopecia
6. Patients with myelodysplastic syndrome/acute myeloid leukaemia
7. Immuno-compromised patients e.g., Human Immunodeficiency Virus (HIV) requiring treatment or active Hepatitis B or C
8. Patients with symptomatic uncontrolled brain metastases. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease (SD) for 28 days
9. Patients considered to be at a high medical risk due to a serious, uncontrolled medical disorder, systemic disease or active, uncontrolled infection
10. Currently pregnant (confirmed with a positive pregnancy test) or breastfeeding.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, Doctor of Medicine, Principal Investigator — Istituto Nazionale Tumori Fondazione G. Pascale, 80131, Napoli, Italy
Locations (46):
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
- Italy (4):
  - Research Site, Bari
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Perugia
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Kielce
  - Research Site, Poznan
- Spain (9):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, San Cristóbal de La Laguna
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- United Kingdom (12):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Newcastle upon Tyne
  - Research Site, Oxford
  - Research Site, Swansea
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00012&attachmentIdentifier=17120550-7e5c-4a45-b05e-ad52fb65aab0&fileName=D0816C00012-SAP-ed5_Final_Redacted.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00012&attachmentIdentifier=4dc4c1bf-d982-4b95-a291-060c8a5e1633&fileName=D0816C00012-CSP-v3_Final_Redacted.pdf&versionIdentifier=
- See also: Synopsis_Primary — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00012&attachmentIdentifier=71181818-9e35-43f9-b5a0-b802bb6b1488&fileName=D0816c00012-synopsis_Primary_Analysis_Redacted_Final_PDFA.pdf&versionIdentifier=
- See also: Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00012&attachmentIdentifier=3988fabf-e95e-41ed-a348-aff3f5a86620&fileName=D0816c00012-synopsis_Redacted_Final_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 8 countries in patients with platinum sensitive relapsed high grade epithelial ovarian (including fallopian tube or primary peritoneal) cancer, who were in complete or partial response to platinum-based chemotherapy.
Pre-assignment Details: 181 patients enrolled and assigned to olaparib: 145 with breast cancer susceptibility gene mutation (BRCAm) status (87 with germline mutations [gBRCAm], 55 with somatic mutations [sBRCAm] and 3 with undetermined BRCAm status), 33 with BRCA-independent homologous recombination repair mutation (HRRm^) status, and 3 enrolled in error (unassigned).
Groups:
- Overall BRCAm: Patients received olaparib capsules orally 400 milligrams (mg) twice daily. Patients in this cohort had BRCAm status, comprising of those with sBRCAm or gBRCAm disease, as well as any patients where the germline or somatic BRCA mutation status was not determined.
- HRRm^: Patients received olaparib capsules orally 400 mg twice daily. Patients in this exploratory cohort had a qualifying mutation in any of the 13 genes involved in the HRR pathway (excluding BRCA1 and BRCA2) (i.e. BRCA-independent HRRm^).
- Unassigned (Not BRCAm, Not HRRm^): Patients received olaparib capsules orally 400 mg twice daily. Patients in this cohort were not classified as being a part of either the BRCAm group or the HRRm^ group and were enrolled in error.
Period: Overall Study
Arm/Group | Overall BRCAm | HRRm^ | Unassigned (Not BRCAm, Not HRRm^)
Started (Enrolled and included in the full analysis set (FAS)) | 145 | 33 | 3
Received Treatment | 143 | 32 | 2
Completed | 50 | 15 | 0
Not Completed | 95 | 18 | 3
Not completed — Other | 0 | 2 | 0
Not completed — Lost to Follow-up | 10 | 0 | 1
Not completed — Death | 48 | 8 | 1
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 1
Not completed — Patient decision | 37 | 8 | 0

BASELINE CHARACTERISTICS:
Population: All patients in the FAS (enrolled and assigned olaparib) were included in the baseline analysis. Where a patient did not meet all the eligibility criteria but was enrolled in error, they were still a part of the FAS.
Groups:
- Overall BRCAm: Patients received olaparib capsules orally 400 mg twice daily. Patients in this cohort had BRCAm status, comprising of those with sBRCAm or gBRCAm disease, as well as any patients where the germline or somatic BRCA mutation status was not determined.
- Total: Total of all reporting groups
Arm/Group | Overall BRCAm | HRRm^ | Unassigned (Not BRCAm, Not HRRm^) | Total
Number analyzed (Participants) | 145 | 33 | 3 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Mean age was calculated for patients with non-missing data (n=164). Only year of birth was reported for 17 patients in the FAS, and consequently, age at enrolment was not imputed for these patients.
  years
    number analyzed (Participants) | 130 | 31 | 3 | 164
    (all) | 60.1 (10.75) | 62.2 (9.74) | 58.7 (9.07) | 60.5 (10.52)
Age, Customized [Count of Participants; unit: Participants] — Population: Age was summarised for patients with non-missing data (n=164). Only year of birth was reported for 17 patients inthe FAS, and consequently, age at enrolment was not imputed for these patients.
  Participants
    number analyzed (Participants) | 130 | 31 | 3 | 164
    <35 years | 0 | 0 | 0 | 0
    ≥35 to <50 years | 27 | 3 | 0 | 30
    ≥50 to <65 years | 54 | 13 | 2 | 69
    ≥65 to <80 years | 48 | 15 | 1 | 64
    ≥80 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 33 | 3 | 181
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 142 | 31 | 3 | 176
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 142 | 31 | 3 | 176
  Asian | 2 | 1 | 0 | 3
  Other | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of PFS. The PFS was defined as the time from the date of enrolment until date of objective radiological disease progression (assessed by the Investigator via Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1]), or death (by any cause in absence of disease progression) regardless of whether the patient withdrew from therapy or received another anti-cancer therapy prior to disease progression. Objective progression was defined as at least a 20% increase in the sum of the diameters of the target lesions (compared to previous minimum sum) and an absolute increase of > 5 millimeters, or an overall non-target lesion assessment of progression or a new lesion. The data cut-off (DCO) for the primary analysis of the study occurred after approximately 60% maturity of PFS in the sBRCAm and all BRCAm patient populations.
Time Frame: Tumour assessments at baseline then every 12 weeks relative to date of enrolment until RECIST 1.1-defined progression. Assessed until primary analysis DCO of 17 April 2020 (up to maximum of 55 months).
Population: The FAS included all enrolled patients who were assigned olaparib. The primary endpoint results for PFS assessment included only BRCAm and sBRCAm patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- sBRCAm: Patients received olaparib capsules orally 400 mg twice daily. Patients in this cohort had sBRCAm disease (i.e. confirmed somatic mutation).
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 18.0 [14.3 to 22.1] | 16.6 [12.4 to 22.2]

2. Secondary Outcome: Overall Survival (OS); Assessed at Primary Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of OS. The OS was defined as the time from the date of enrolment until death due to any cause regardless of whether the patient withdrew from therapy or received another anti-cancer therapy. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Pre-specified analysis of OS was performed at the time of primary analysis of PFS; a further analysis of OS was performed after approximately 60% maturity of OS in the sBRCAm and all BRCAm patient populations (and reported as a separate outcome measure).
Time Frame: From baseline until death due to any cause. Assessed until primary analysis DCO of 17 April 2020 (up to maximum of 55 months).
Population: The FAS included all enrolled patients who were assigned olaparib. The secondary endpoint results for OS assessment included only BRCAm and sBRCAm patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Overall BRCAm: Patients received olaparib capsules orally 400 mg twice daily. Patients in this cohort had BRCAm status, comprising of those with sBRCAm or gBRCAm disease, as well as any patients where the germline or somatic BRCA mutation status was not confirmed.
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 47.6 [36.1 to NA] — The upper limit 95% confidence interval (CI) could not be calculated as it was not reached. | NA [33.2 to NA] — The median and upper limit 95% CI could not be calculated as they were not reached.

3. Secondary Outcome: Time to Second Progression (PFS2) or Death; Assessed at Primary Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of PFS2. The PFS2 was defined as the time from the date of enrolment to the earliest progression event subsequent to that used for the primary variable PFS or death (by any cause) in the absence of progression. Patients whose progression event for PFS was death had this counted as a progression event for PFS2 also. The date of second progression was recorded by the Investigator and defined according to local standard clinical practice and could involve any of the following: objective radiological, symptomatic, cancer antigen-125 (CA-125) progression or death. Pre-specified analysis of PFS2 was performed at the time of the primary analysis; a further analysis of PFS2 was performed at the final analysis (and reported as a separate outcome measure).
Time Frame: Tumour assessments (and blood samples for CA-125, if applicable) at baseline then every 12 weeks relative to date of enrolment until second progression. Assessed until primary analysis DCO of 17 April 2020 (up to maximum of 55 months).
Population: The FAS included all enrolled patients who were assigned olaparib. The secondary endpoint results for PFS2 assessment included only BRCAm and sBRCAm patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 30.9 [24.7 to 40.0] | 24.7 [21.8 to 36.1]

4. Secondary Outcome: Time to First Subsequent Therapy (Treatment) or Death (TFST); Assessed at Primary Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of TFST. The TFST was defined as the time from the date of enrolment to the earlier of first subsequent anti-cancer therapy start date (excluding radiotherapy), or death date. Pre-specified analysis of TFST was performed at the time of the primary analysis; a further analysis of TFST was performed at the final analysis (and reported as a separate outcome measure).
Time Frame: From enrolment to first subsequent therapy or death. Assessed every 12 weeks following treatment discontinuation. Assessed until primary analysis DCO of 17 April 2020 (up to maximum of 55 months).
Population: The FAS included all enrolled patients who were assigned olaparib. The secondary endpoint results for TFST assessment included only BRCAm and sBRCAm patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 37.6 [23.5 to 47.6] | 31.5 [19.5 to NA] — The upper limit 95% CI could not be calculated as it was not reached.

5. Secondary Outcome: Time to Second Subsequent Therapy (Treatment) or Death (TSST); Assessed at Primary Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of TSST. The TSST was defined as the time from the date of enrolment to the earlier of the date of second subsequent anti-cancer therapy start date, or death date. Pre-specified analysis of TSST was performed at the time of the primary analysis; a further analysis of TSST was performed at the final analysis (and reported as a separate outcome measure).
Time Frame: From enrolment to second subsequent therapy or death. Assessed every 12 weeks following treatment discontinuation. Assessed until primary analysis DCO of 17 April 2020 (up to maximum of 55 months).
Population: The FAS included all enrolled patients who were assigned olaparib. The secondary endpoint results for TSST assessment included only BRCAm and sBRCAm patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 47.6 [29.4 to NA] — The upper limit 95% CI could not be calculated as it was not reached. | NA [24.7 to NA] — The median and upper limit 95% CI could not be calculated as they were not reached.

6. Secondary Outcome: Time to Discontinuation of Treatment or Death (TDT)
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of TDT. The TDT was defined as the time from the date of enrolment to the earlier of the date of study treatment discontinuation or death.
Time Frame: From enrolment to study treatment discontinuation or death (up to maximum of 6 years).
Population: The FAS included all enrolled patients who were assigned olaparib. The secondary endpoint results for TDT assessment included only BRCAm and sBRCAm patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 19.8 [14.3 to 22.9] | 19.0 [13.5 to 22.8]

7. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Ovarian (FACT-O) Trial Outcome Index (TOI) Scores Over Time
Description: To assess the Quality of Life (QoL) of patients with BRCAm and sBRCAm ovarian cancer by evaluation of FACT-O TOI. The TOI score was derived from the sum of the scores of the 25 items included in the physical well-being (7 items), functional well-being (7 items), and additional concerns ovarian cancer subscale (11 items) of the FACT-O questionnaire version 4. The FACT-O TOI score ranges from 0-100, with a higher score indicating better QoL. A change (increase or decrease) in score of at least 10 points from baseline was defined as clinically meaningful. A positive change in score from baseline indicates an improvement.
Time Frame: QoL questionnaires at baseline, Day 29 (Week 4), then every 12 weeks for 24 months or DCO for primary analysis, whichever came first. QoL questionnaires also collected at discontinuation of study treatment visit and 30 days post last dose.
Population: The FAS-FACT-O-TOI population included all enrolled patients who were assigned olaparib excluding patients who did not have FACT-O TOI score at baseline and patients who did not have any FACT-O TOI score post-baseline. The secondary endpoint results for FACT-O TOI assessment included only BRCAm and sBRCAm patients.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 131 | 50
scores on a scale
  Week 4: number analyzed (Participants) | 126 | 47
  Week 4 | -2.2 (9.82) | -1.9 (9.59)
  Week 16: number analyzed (Participants) | 91 | 31
  Week 16 | -1.3 (10.04) | -0.3 (10.85)
  Week 28: number analyzed (Participants) | 82 | 30
  Week 28 | 1.2 (9.44) | 3.2 (10.25)
  Week 40: number analyzed (Participants) | 80 | 28
  Week 40 | 1.6 (10.72) | 4.1 (10.48)
  Week 52: number analyzed (Participants) | 70 | 24
  Week 52 | 3.2 (9.03) | 4.9 (7.84)
  Week 64: number analyzed (Participants) | 60 | 23
  Week 64 | 1.8 (9.88) | 0.8 (9.72)
  Week 76: number analyzed (Participants) | 57 | 20
  Week 76 | 1.4 (9.27) | 0.3 (9.83)
  Week 88: number analyzed (Participants) | 46 | 15
  Week 88 | 2.0 (9.97) | 1.5 (10.86)
  Week 100: number analyzed (Participants) | 34 | 11
  Week 100 | -0.2 (9.41) | -3.5 (7.54)
  Discontinuation of olaparib visit: number analyzed (Participants) | 36 | 16
  Discontinuation of olaparib visit | -4.7 (13.00) | -7.4 (15.53)
  30 days post discontinuation: number analyzed (Participants) | 52 | 24
  30 days post discontinuation | -8.0 (13.45) | -4.3 (13.36)

8. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Total Scores Over Time
Description: To assess the QoL of patients with BRCAm and sBRCAm ovarian cancer by evaluation of FACIT-F. The FACIT-F is a 13-item questionnaire to assess patients' fatigue experience and its impact on their daily lives over the past 7 days. The FACIT-F total score ranges from 0-52, with a higher score indicating a lower level of fatigue (and better QoL). Changes in scores of ≥3 points were defined to be clinically meaningful. A positive change in score from baseline indicates an improvement.
Time Frame: as for outcome 7
Population: The FAS-FACIT-F population included all enrolled patients who were assigned olaparib excluding patients who did not have FACIT-F total score at baseline and patients who did not have any FACIT-F total score post-baseline. The secondary endpoint results for FACIT-F assessment included only BRCAm and sBRCAm patients.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 136 | 53
scores on a scale
  Week 4: number analyzed (Participants) | 130 | 48
  Week 4 | -2.9 (8.21) | -2.9 (7.58)
  Week 16: number analyzed (Participants) | 95 | 34
  Week 16 | -2.5 (7.54) | -2.7 (9.26)
  Week 28: number analyzed (Participants) | 83 | 31
  Week 28 | -1.2 (7.95) | -0.6 (7.25)
  Week 40: number analyzed (Participants) | 83 | 31
  Week 40 | -0.3 (7.91) | 0.9 (7.02)
  Week 52: number analyzed (Participants) | 76 | 29
  Week 52 | 0.6 (7.43) | 1.3 (7.25)
  Week 64: number analyzed (Participants) | 65 | 25
  Week 64 | 0.8 (7.26) | 0.5 (8.47)
  Week 76: number analyzed (Participants) | 58 | 21
  Week 76 | -0.3 (8.57) | -1.1 (8.74)
  Week 88: number analyzed (Participants) | 46 | 14
  Week 88 | 0.3 (8.45) | -0.9 (5.81)
  Week 100: number analyzed (Participants) | 34 | 11
  Week 100 | -0.4 (8.59) | -1.3 (8.75)
  Discontinuation of olaparib visit: number analyzed (Participants) | 37 | 16
  Discontinuation of olaparib visit | -2.3 (9.01) | -2.7 (9.32)
  30 days post discontinuation: number analyzed (Participants) | 53 | 24
  30 days post discontinuation | -5.2 (11.16) | -3.8 (9.65)

9. Secondary Outcome: Change From Baseline in Functional Living Index-Emesis (FLIE) Questionnaire Total Scores Over Time
Description: The FLIE captures the impact of nausea and vomiting on patient's QoL. The FLIE consists of 18 items (9 nausea-specific and 9 vomiting-specific items), rated from 1 to 7. Two domain scores and a total score are derived; the total score ranges 18-126 and a higher score indicates a lower impact (and better QoL). A positive change in score from baseline indicates an improvement.
Time Frame: FLIE questionnaires at baseline, weekly until Day 29 (Week 4), then every 12 weeks for 24 months or DCO for primary analysis, whichever came first. FLIE questionnaires also collected at discontinuation of study treatment visit and 30 days post last dose.
Population: The FAS-FLIE population included all enrolled patients who were assigned olaparib excluding patients who did not have FLIE total score at baseline and patients who did not have any FLIE total score post-baseline. The secondary endpoint results for FLIE assessment included only BRCAm and sBRCAm patients.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 114 | 46
scores on a scale
  Week 1: number analyzed (Participants) | 105 | 42
  Week 1 | -6.1 (18.62) | -1.6 (18.28)
  Week 2: number analyzed (Participants) | 101 | 39
  Week 2 | -4.5 (18.40) | -2.6 (15.97)
  Week 3: number analyzed (Participants) | 102 | 40
  Week 3 | -4.1 (14.57) | -3.9 (13.23)
  Week 4: number analyzed (Participants) | 103 | 39
  Week 4 | -4.8 (18.48) | -5.4 (19.92)
  Week 16: number analyzed (Participants) | 80 | 29
  Week 16 | -2.3 (11.50) | -6.3 (11.00)
  Week 28: number analyzed (Participants) | 73 | 28
  Week 28 | -1.6 (13.87) | -3.0 (7.94)
  Week 40: number analyzed (Participants) | 72 | 28
  Week 40 | -0.1 (14.07) | -3.2 (14.56)
  Week 52: number analyzed (Participants) | 64 | 26
  Week 52 | 0.9 (14.41) | -1.9 (11.64)
  Week 64: number analyzed (Participants) | 54 | 23
  Week 64 | -0.2 (15.93) | -1.0 (20.77)
  Week 76: number analyzed (Participants) | 49 | 19
  Week 76 | 0.9 (14.14) | 0.6 (6.60)
  Week 88: number analyzed (Participants) | 42 | 14
  Week 88 | 2.2 (10.04) | -1.3 (9.29)
  Week 100: number analyzed (Participants) | 32 | 11
  Week 100 | 0.4 (10.37) | 0.1 (13.19)
  Discontinuation of olaparib visit: number analyzed (Participants) | 28 | 12
  Discontinuation of olaparib visit | -0.7 (20.17) | -8.8 (21.57)
  30 days post discontinuation: number analyzed (Participants) | 39 | 18
  30 days post discontinuation | -5.2 (17.02) | -5.6 (15.69)

10. Secondary Outcome: OS; Assessed at Final Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of OS. The OS was defined as the time from the date of enrolment until death due to any cause regardless of whether the patient withdrew from therapy or received another anti-cancer therapy. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive.
Time Frame: From baseline until death due to any cause (up to maximum of 6 years).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 46.8 [37.9 to 54.4] | 43.2 [31.7 to NA] — The upper limit 95% CI could not be calculated as it was not reached.

11. Secondary Outcome: PFS2 or Death; Assessed at Final Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of PFS2. The PFS2 was defined as the time from the date of enrolment to the earliest progression event subsequent to that used for the primary variable PFS or death (by any cause) in the absence of progression. Patients whose progression event for PFS was death had this counted as a progression event for PFS2 also. The date of second progression was recorded by the Investigator and defined according to local standard clinical practice and could involve any of the following: objective radiological, symptomatic, CA-125 progression or death.
Time Frame: Tumour assessments (and blood samples for CA-125, if applicable) at baseline then every 12 weeks relative to date of enrolment until second progression (up to maximum of 6 years).
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 34.0 [29.3 to 44.2] | 29.3 [23.7 to 44.2]

12. Secondary Outcome: TFST; Assessed at Final Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of TFST. The TFST was defined as the time from the date of enrolment to the earlier of first subsequent anti-cancer therapy start date (excluding radiotherapy), or death date.
Time Frame: From enrolment to first subsequent therapy or death. Assessed every 12 weeks following treatment discontinuation (up to maximum of 6 years).
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 32.1 [25.8 to 40.0] | 31.7 [18.0 to NA] — The upper limit 95% CI could not be calculated as it was not reached.

13. Secondary Outcome: TSST; Assessed at Final Analysis
Description: To assess the real-world clinical effectiveness of olaparib maintenance monotherapy in patients with BRCAm and sBRCAm ovarian cancer by assessment of TSST. The TSST was defined as the time from the date of enrolment to the earlier of the date of second subsequent anti-cancer therapy start date, or death date.
Time Frame: From enrolment to second subsequent therapy or death. Assessed every 12 weeks following treatment discontinuation (up to maximum of 6 years).
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall BRCAm | sBRCAm
Number analyzed (Participants) | 145 | 55
months | 38.4 [31.5 to NA] — The upper limit 95% CI could not be calculated as it was not reached. | 32.1 [25.8 to 44.7]

ADVERSE EVENTS:
Time Frame: From first dose of olaparib up to and including 30 days following the date of discontinuation of olaparib. Maximum timeframe of approximately 6 years.
Description: Adverse events are reported for the safety analysis set which included all patients who received at least one dose of olaparib. All- cause mortality was determined for patients in the FAS (enrolled and assigned olaparib).
Groups:
- gBRCAm: Patients received olaparib capsules orally 400 mg twice daily. Patients in this cohort had gBRCAm disease (i.e. confirmed germline mutation).
- HRRm: Patients received olaparib capsules orally 400 mg twice daily. Patients in this exploratory cohort had a qualifying mutation in any of the 13 genes involved in the HRR pathway (excluding BRCA1 and BRCA2) (i.e. BRCA-independent HRRm^).
Arm/Group | gBRCAm | sBRCAm | Overall BRCAm | HRRm | Unassigned (Not BRCAm, Not HRRm^)
All-Cause Mortality (participants affected / at risk) | 40/87 | 28/55 | 68/145 | 14/33 | 2/3
Serious Adverse Events (participants affected / at risk) | 27/87 | 13/55 | 40/143 | 7/32 | 1/2
Other Adverse Events (participants affected / at risk) | 79/87 | 51/55 | 131/143 | 29/32 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gBRCAm (N=87) | sBRCAm (N=55) | Overall BRCAm (N=143) | HRRm (N=32) | Unassigned (Not BRCAm, Not HRRm^) (N=2)
Anaemia (Blood and lymphatic system disorders) | 7 (10) | 5 (6) | 12 (16) | 1 (10) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gBRCAm (N=87) | sBRCAm (N=55) | Overall BRCAm (N=143) | HRRm (N=32) | Unassigned (Not BRCAm, Not HRRm^) (N=2)
Anaemia (Blood and lymphatic system disorders) | 38 (55) | 19 (31) | 57 (86) | 11 (16) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 8 (8) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 12 (16) | 4 (10) | 16 (26) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 6 (7) | 11 (12) | 1 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 2 (2) | 8 (9) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 12 (20) | 23 (31) | 8 (9) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 3 (4) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (13) | 4 (6) | 13 (19) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 8 (9) | 13 (15) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (16) | 9 (11) | 24 (27) | 8 (9) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (5) | 0 (0) | 3 (5) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 49 (86) | 28 (36) | 78 (123) | 19 (30) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (41) | 14 (27) | 38 (68) | 10 (25) | 1 (1)
Asthenia (General disorders) | 13 (19) | 11 (14) | 24 (33) | 2 (2) | 0 (0)
Fatigue (General disorders) | 38 (46) | 22 (25) | 60 (71) | 15 (18) | 1 (1)
Influenza like illness (General disorders) | 7 (8) | 2 (2) | 9 (10) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 5 (6) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 7 (13) | 0 (0) | 7 (13) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (12) | 3 (4) | 12 (16) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 6 (6) | 8 (9) | 1 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (9) | 6 (13) | 11 (22) | 4 (6) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (11) | 1 (1) | 8 (12) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 8 (21) | 3 (3) | 11 (24) | 4 (6) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 3 (5) | 5 (7) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (8) | 2 (3) | 7 (11) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 5 (6) | 1 (1) | 6 (7) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 5 (14) | 2 (7) | 7 (21) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 7 (8) | 17 (18) | 5 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (11) | 4 (4) | 11 (15) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6) | 9 (10) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 5 (6) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2) | 6 (9) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 13 (21) | 2 (3) | 15 (24) | 5 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 8 (10) | 3 (3) | 11 (13) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 11 (16) | 3 (11) | 14 (27) | 6 (8) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 3 (3) | 7 (7) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 3 (3) | 7 (7) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (4) | 11 (11) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 14 (27) | 8 (10) | 23 (38) | 5 (5) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 6 (8) | 6 (8) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 5 (5) | 2 (3) | 7 (8) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 2 (4) | 8 (13) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (20) | 2 (2) | 8 (22) | 2 (3) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 6 (8) | 17 (23) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 5 (5) | 14 (17) | 6 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (25) | 4 (8) | 13 (33) | 6 (7) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 4 (6) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (9) | 4 (4) | 11 (13) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 7 (8) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 6 (6) | 3 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 6 (6) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02476968/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02476968/SAP_001.pdf